CLINICAL TRIAL: NCT05876884
Title: Efficacy of a Low-cost Warming Mattress Celsi Warmer for the Management of Hypothermic Newborns at Muhimbili National Hospital, Dar es Salaam, Tanzania
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: William Marsh Rice University (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); Ifakara Health Institute (Other); Ministry of Health, Community Development, Gender, Elderly, and Children (MOHCDGEC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TZ Celsi Warmer
Record Dates: First submitted 2023-04-03; First posted 2023-05-26 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Neonatal Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypothermic Neonates (90) (Experimental): Any neonate who been identified as in need of thermal care defined as having a moderate hypothermic temperature (32.0 - 36.0°C) as the last temperature recorded in hospital chart, or during recruitment procedures will be placed on the Celsi Warmer mattress
  Interventions: Device: Celsi Warmer Mattress

INTERVENTIONS:
Device: Celsi Warmer Mattress — The hypothermic neonate will be placed on the Celsi Warmer mattress and a temperature probe will be placed on the neonate to monitor the temperature of the neonate for up to 24 hours of intervention time

SUMMARY:
The prevalence of hypothermia across low-resource settings is high, especially in countries with high neonatal mortality rates. If left untreated, hypothermia can additionally result in a significant comorbidity, and has been linked to a reduction in the effectiveness of treatment for other newborn conditions. Thermal care for hypothermic newborns is not widely available in low-resource settings due to cost, and lack of consumables and spare parts. In this study, the research team will evaluate the efficacy of a novel neonatal warming mattress intreating hypothermic newborns. The warming mattress, 'Celsi Warmer', has been developed by Rice360 Institute for Global Health Technologies, in conjunction with African clinicians, to be a robust, low-cost, and easy-to-use warming mattress which can address the challenges of hypothermia. This is a single-arm, non-randomized, prospective intervention study. Up to90eligible infants at Muhimbili National Hospital (MNH) at Upanga Neonatal Unit will be recruited to evaluate the efficacy of Celsi Warmer in rewarming hypothermic newborns. Infants temperature will be monitored during thermal intervention and the performance of the device will be evaluated. The temperatures of each infant will be compared before, during, and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

Any neonate who:

1. Is currently being treated at study location
2. Is an inborn admission to the neonatal ward
3. Whose parents or guardians provided a written informed consent
4. Whose parents or guardians providing informed consent are 18 years old or older
5. Has a current weight of greater than or equal to 1.0 kg and less than or equal to 4.0kg
6. Has been identified as in need of thermal care defined as having a moderate hypothermic temperature (32.0-36.0°C) as the last temperature recorded in hospital chart, or during recruitment procedures; and
7. Is unable to be enrolled in Kangaroo Mother Care (KMC) for reasons including, but not limited to: a.Mother/guardian unable or unavailable to provide KMC b.Under observation in NICU before transfer to KMC c.No space in KMC d.Clinician's discretion
8. May be receiving other medical treatments, including but not limited to, CPAP, oxygen therapy, IV fluids, management and monitoring of common newborn conditions such as hypoglycemia, and/or hyperbilirubinemia via LED phototherapy

The study will not interfere with any other treatment being provided at the ward, and it will not delay the participant from transferring to KMC or being discharged

Exclusion Criteria:

Any neonate who:

1. Requires mechanical ventilation
2. Is deemed in need of intensive care by the hospital staff who is providing care,including but not limited to: a.neonates with severe anemia and/or any suspected hematological disorders, and/or b. Neonates with obvious congenital anomalies, and/or c.neonates suspected with hypo/hyperthyroidism or any hormonal disorders
3. Has been diagnosed with birth asphyxia
4. Presents a condition that precludes the use of the temperature sensor and/or abdominal belt including but not limited to, gastroschisis, known umbilical cord infection, known skin infection
5. Whose clinician presents concerns about their participation
6. Is receiving treatment that participation in the study would interfere with, i.e.transferring to KMC

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Broad Objective | 1 year
  To evaluate the clinical efficacy and safety of the Celsi Warmer in rewarming hypothermic newborns by comparing the Celsi Warmer's accuracy in measuring neonatal temperature compared to the gold standard, axillary temperature readings.

SECONDARY OUTCOMES:
Efficacy of the Device | 1 year
  To assess the performance of the Celsi Warmer in rewarming hypothermic newborns by measuring the incidence of attainment of normothermia (36.5-37.5°C)
Safety of Device | 1 year
  To measure the infant's rate of temperature (°C) increase through thermoregulatory intervention.
Safety of Device | 1 year
  To evaluate the local effect of the abdominal belt on newborn's skin by looking at any evidence of skin irritation
Safety of Device | 1 year
  To evaluate any incidence of hyperthermia (>37.5°C) during the thermoregulation intervention.
Safety of Device | 1 year
  To report any incidence of rebound hypothermia ( < 36.5°C) (post-intervention hypothermia) up to 72 hours from the initial encounter

CONTACTS AND LOCATIONS:
Locations (1):
- Muhimbili National Hospital, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No